CLINICAL TRIAL: NCT06715319
Title: A Double-blind, Randomized Phase 3 Trial Evaluating the Efficacy and Safety of Obecholic Acid Versus Placebo, in Combination with Ursodeoxycholic Acid in Primary Biliary Cirrhosis Patients with an Inadequate Response to Ursodeoxycholic Acid
Brief Title: Obeticholic Acid Versus Placebo, in Combination with Ursodeoxycholic Acid in Patients with Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDZJ-OCA-202011
Record Dates: First submitted 2024-11-27; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: PBC
MeSH Terms: interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCA and UDCA (Experimental): OCA 5 mg once daily for 3 months and then titrating up to 10 mg based on tolerability and response.
  Subjects receiving UDCA continued taking UDCA throughout the trial. If the subjects could not tolerate UDCA, they were not treated with UDCA.
  Interventions: Drug: OCA; Drug: UDCA
- Placebo and UDCA (Placebo Comparator): Placebo once daily. Subjects receiving UDCA continued taking UDCA throughout the trial.
  Interventions: Drug: UDCA; Drug: Placebo

INTERVENTIONS:
Drug: OCA — OCA 5 mg once daily in combination with UDCA for 12 weeks and then titrating up to 10 mg based on tolerability and response for remainder of double-blind period.
  Other Names: Obeticholic Acid
  Arms: OCA and UDCA
Drug: UDCA — 13~15 mg/kg/day
Drug: Placebo — Once a day (QD) by mouth (PO)
  Arms: Placebo and UDCA

SUMMARY:
This is a Phase III, randomized, double-blind, multicentre study assessing the efficacy and safety of obecholic acid and Ursodeoxycholic Acid(UDCA) compared with placebo and UDCA in treating of primary biliary cirrhosis (PBC) in adults with an inadequate response to UDCA.

DETAILED DESCRIPTION:
The main objectives of the study were to assess the effects of Obeticholic Acid (OCA) on serum alkaline phosphatase (ALP) and total bilirubin, together as a composite endpoint and on safety in participants with PBC.

The study included 2 phases: a 6-month randomized, double-blind (DB), placebo-controlled, parallel-group phase, followed by a 6-month DB treatment phase. In the 6-month randomized, DB placebo-controlled phase, patients will receive OCA/placebo with a dosage of 5 mg once daily for the first 3 months. After the first 3 months, for patients who have not achieved an adequate reduction in ALP and/or total bilirubin and who are tolerating OCALIVA/placebo, increase to a maximum dosage of 10 mg once daily.

Participants in the 6-month DB treatment phase were eligible to receive the treatment of OCA, especially those who received placebo, for patients who have not achieved an adequate reduction in ALP and/or total bilirubin, will receive OCA with a dosage of 5 mg once daily for the first 3 months. After the first 3 months, for patients who have not achieved an adequate reduction in ALP and/or total bilirubin and who are tolerating OCALIVA, increase to a maximum dosage of 10 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Definite PBC diagnosis, as demonstrated by the presence of ≥ 2 of the following 3 diagnostic factors: ① Indicators reflecting cholestasis such as elevated ALP；② Positive antimitochondrial antibody (AMA) or AMA-M2, or positive PBC-specific antibody (anti-GP210 and/or anti-SP100) if AMA negative；③ Liver biopsy consistent with PBC;
2. At least 1 of the following qualifying biochemistry values: ① ALP ≥ 1.67x ULN；② Total bilirubin > ULN but < 2x ULN；
3. Taking UDCA for at least 6 months (stable dose for ≥ 2 months) prior to the first dose；
4. Patients of childbearing potential must agree to take contraception during the study and for 1 month after the last day of treatment;
5. Patients capable of giving written informed consent.

Exclusion Criteria:

1. History or presence of other concomitant liver diseases including:

   Hepatitis C virus (HCV) infection; participants with active hepatitis B (HBV) infection will be excluded, however, participants who have seroconverted (hepatitis B surface antigen [Hbs Ag] and hepatitis B e antigen [Hbe Ag] negative) may be included after consultation with the medical monitor.

   Primary sclerosing cholangitis (PSC) Alcoholic liver disease Definite autoimmune liver disease or overlap hepatitis Nonalcoholic steatohepatitis (NASH) Gilbert's Syndrome (due to interpretability of bilirubin levels)Child-pugh grade B or C
2. Presence of clinical complications of PBC or clinically significant hepatic decompensation, including:

   History of liver transplantation, current placement on a liver transplant list or current Model for End Stage Liver Disease (MELD) score ≥ 15 Portal hypertension with complications, including: known gastric or large esophageal varices, poorly controlled or diuretic resistant ascites, history of variceal bleeds or related therapeutic or prophylactic interventions (for example, beta blockers, insertion of variceal bands or transjugular intrahepatic portosystemic shunt [TIPS]), or hepatic encephalopathy Cirrhosis with complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma, bilirubin > 2x ULN Hepatorenal syndrome (type I or II) or Screening serum creatinine > 2 mg/deciliter dL) (178 micromoles [µmol])/liter [L])
3. Participants with severe pruritus or those requiring systemic treatment for pruritus (for example, with bile acid sequestrants [BAS] or rifampicin) within 2 months prior to the first dose
4. Patients who took obeticholic acid within 3 months prior to the first dose
5. Administration of the following drugs within 1 month prior to the first dose: azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate mofetil, pentoxifylline, bicyclol and with S.chinensis ingredients; fenofibrate or other fibrates; budesonide and other systemic corticosteroids; hepatotoxic drugs (including α-methyldopa, sodium valproate, isoniazid, nitrofurantoin, etc.);
6. Administration of the following drugs within 2 months prior to the first dose: antibodies or immunotherapy against interleukins or other cytokines or chemokines.
7. ALT≥ 10 × ULN with/or ALT≥ 10 × ULN;
8. Direct bilirubin>3×ULN;
9. Serum creatinine (Cr) ≥ 1.5 × ULN and serum creatinine clearance < 60 mL/min;
10. History or presence of clinically concerning cardiac arrhythmias likely to affect survival during the trial, or prolongation of Screening (pretreatment) QT or QTc interval;
11. Women who are pregnant or lactating;
12. Known history of human immunodeficiency virus (HIV) infection
13. Presence of any other disease or condition that is interfering with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the intestine. Participants with inflammatory bowel disease or who have undergone gastric bypass procedures will be excluded (gastric lap band is acceptable)
14. Medical conditions that may cause nonhepatic increases in ALP (for example, Paget's disease) or which may diminish life expectancy to < 2 years, including known cancers (except carcinomas in situ or other stable, relatively benign conditions such as chronic lymphatic leukemia)
15. Other clinically significant medical conditions that are not well controlled or for which medication needs are anticipated to change during the trial;
16. Anticipated changes to current concomitant medications during the trial;
17. Mental instability or incompetence;
18. Other circumstances that are deemed not appropriate for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint Alkaline Phosphatase (ALP) And Total Bilirubin | up to 6 months
  Composite Endpoint : Percentage of participants at Month 12 with ALP < 1.67 x upper limit of normal (ULN) and total bilirubin ≤ ULN and ALP decrease of ≥ 15% from baseline.

SECONDARY OUTCOMES:
Percentage of PBC patients reaching the composite endpoint after 12 weeks, 36 weeks and 48 weeks of treatment | up to 12 months
  Composite Endpoint : Percentage of participants at Month 12 with ALP < 1.67 x upper limit of normal (ULN) and total bilirubin ≤ ULN and ALP decrease of ≥ 15% from baseline.
Absolute change and percentage change of ALP from baseline to Month 3, 6, 9 and 12 | up to 12 months
  Blood samples were evaluated for ALP from baseline to Month 3, 6, 9 and 12 are presented.
Absolute change and percentage change of total bilirubin from baseline to Month 3, 6, 9 and 12 | up to 12 months
  Blood samples were evaluated for total bilirubin from baseline to Month 3, 6, 9 and 12 are presented.
Absolute change and percentage change of direct bilirubin from baseline to Month 3, 6, 9 and 12 | up to 12 months
  Blood samples were evaluated for direct bilirubin from baseline to Month 3, 6, 9 and 12 are presented.
Absolute change and percentage change of alanine transaminase(ALT) from baseline to Month 3, 6, 9 and 12 | up to 12 months
  Blood samples were evaluated for ALT from baseline to Month 3, 6, 9 and 12 are presented.
Absolute change and percentage change of alkaline phosphatase(AST) from baseline to Month 3, 6, 9 and 12 | up to 12 months
  Blood samples were evaluated for AST from baseline to Month 3, 6, 9 and 12 are presented.
Absolute change and percentage change of gamma glutamyl transpeptidase(GGT) from baseline to Month 3, 6, 9 and 12 | up to 12 months
  Blood samples were evaluated for GGT from baseline to Month 3, 6, 9 and 12 are presented.
Incidence of Treatment-Emergent Adverse Events | up to 12 months
  Adverse Events will be evaluated in terms of adverse events (graded by CTCAE version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China